CLINICAL TRIAL: NCT04991350
Title: Comparison of the Effect of Ranibizumab Versus Bevacizumab on the Macular Perfusion in Diabetic Macular Edema Using OCTA
Brief Title: Effect of Ranibizumab Versus Bevacizumab on the Macular Perfusion in Diabetic Macular Edema
Acronym: REBEL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Gehad Elnahry, Lecturer of Ophthalmology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU372021
Record Dates: First submitted 2021-07-24; First posted 2021-08-05 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Macular Edema; Macular Ischemia; Diabetic Retinopathy; Vascular Endothelial Growth Factor Overexpression
Keywords: Diabetic macular edema; Macular perfusion; Optical coherence tomography angiography; Anti-VEGF
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ranibizumab Group (Active Comparator): Patients will receive monthly ranibizumab injections for 3 months.
  Interventions: Drug: Intravitreal ranibizumab
- Bevacizumab Group (Active Comparator): Patients will receive monthly bevacizumab injections for 3 months.
  Interventions: Drug: Intravitreal bevacizumab

INTERVENTIONS:
Drug: Intravitreal ranibizumab — Intravitreal injection of 0.3 mg/0.05 ml ranibizumab will be performed monthly for 3 months.
  Other Names: Lucentis
  Arms: Ranibizumab Group
Drug: Intravitreal bevacizumab — Intravitreal injection of 1.25 mg/0.05 ml bevacizumab will be performed monthly for 3 months.
  Other Names: Avastin
  Arms: Bevacizumab Group

SUMMARY:
The Early Treatment Diabetic Retinopathy Study (ETDRS) group founded guidelines for treating patients with clinically significant diabetic macular edema (DME) with focal/grid macular laser photocoagulation. Since then, macular laser, and steroids, were the main therapies for the treatment of DME until anti-vascular endothelial growth factors (anti-VEGF) drugs were developed after a growing body of scientific evidence implicated VEGF in the pathophysiologic process of DME.

Anti-VEGF drugs have been implicated in the treatment of DME. VEGF has been shown to play an important role in the occurrence of increased vascular permeability in DME. VEGF levels are significantly higher in patients with DME and extensive leakage than in patients with minimal leakage.

Many studies such as Diabetic Retinopathy Clinical Research [DRCR] Network studies, RESTORE Study, RISE and RIDE Research Group, and The BOLT Study have supported the use of anti-VEGF agents in the treatment of DME with better visual outcomes using anti-VEGF injections alone or in combination with other treatments.

Several ocular complications of intravitreal anti-VEGF injections have been reported including endophthalmitis, cataract, and retinal detachment. The different effects on macular perfusion between different anti-VEGFs have yet to be fully concluded with mixed conclusions that it increases or decreases or has no effect on perfusion of the macula in response to Anti-VEGF treatment. In many of these studies, however, patients with more ischemic retinas were not included. Retinal ischemia is a vital factor determining the diabetic retinopathy progression and prognosis.

Optical coherence tomography angiography (OCTA) detects blood flow by analyzing signal decorrelation between two sequential OCT cross-sectional scans at the same location. As it detects the movements of red blood corpuscles within the vessels, compared to the stationary retinal surroundings, which will result in signal disparity and imaging The split-spectrum amplitude-decorrelation angiography (SSADA) algorithm improves the signal to noise ratio. OCTA is considered a reliable tool in the detection and quantification of macular ischemia in diabetics.

In this study, the investigators aim to compare the effect of repeated intravitreal injections of ranibizumab and bevacizumab on the perfusion of different capillary layers in the macula of diabetic patients using OCTA.

DETAILED DESCRIPTION:
Diabetic retinopathy is the major cause of blindness in developed but also in developing countries. The disruption of the blood-retinal barrier and the subsequent accumulation of fluid in the intraretinal layers result in diabetic macular edema (DME), the leading cause of central vision loss in these patients.

The Early Treatment Diabetic Retinopathy Study (ETDRS) group founded guidelines for treating patients with clinically significant DME (CSME) with focal/grid macular laser photocoagulation. Since then, macular laser, and steroids, were the main therapies for treatment of DME until anti-vascular endothelial growth factors (anti-VEGF) drugs were developed after a growing body of scientific evidence implicated VEGF in the pathophysiologic process of DME.

Anti-VEGF drugs have been implicated in the treatment of DME. VEGF has been shown to play an important role in the occurrence of increased vascular permeability in DME. VEGF levels are significantly higher in patients with DME and extensive leakage than in patients with minimal leakage.

Many studies such as Diabetic Retinopathy Clinical Research [DRCR] Network studies, RESTORE Study, RISE and RIDE Research Group, and The BOLT Study have supported the use of anti-VEGF agents in the treatment of DME with better visual outcomes using anti-VEGF injections alone or in combination with other treatments.

DRCR network protocol T found statistically insignificant difference between ranibizumab and bevacizumab on visual acuity and central macular thickness in diabetic macular edema.

Several ocular complications of intravitreal anti-VEGF injections have been reported including endophthalmitis, cataract, and retinal detachment. The different effects on macular perfusion between different anti-VEGFs have yet to be fully concluded with mixed conclusions that it increases or decreases or has no effect on perfusion of macula in response to Anti-VEGF treatment.in many of these studies, however, patients with more ischemic retinas were not included. Retinal ischemia is a vital factor determining the diabetic retinopathy progression and prognosis.

Using ocular ultrasound some studies showed retinal arteriolar vasoconstriction in eyes treated with anti-VEGF, while others showed decreased blood flow velocities in all retro-bulbar arteries after intravitreal injection of anti-VEGF. This may indicate that anti-VEGF may have an effect on ocular perfusion.

Fluorescein angiography (FA) was the method used to assess changes in macular perfusion after anti-VEGF injections in most of the studies. Despite its clinical value, however, FA is known to have documented risks. Optical coherence tomography angiography (OCTA) is an excellent non-invasive modality to acquire high-resolution images of the retinal vasculature that can be utilized in the treatment of retinal disease without the need for dye injection. It allows the visualization of both the superficial and deep retinal capillary layers separately and the construction of microvascular flow maps.

OCTA detects blood flow by analyzing signal decorrelation between two sequential OCT cross-sectional scans at the same location. As it detects the movements of red blood corpuscles within the vessels, compared to the stationary retinal surroundings, which will result in signal disparity and imaging The split-spectrum amplitude-decorrelation angiography (SSADA) algorithm improves the signal to noise ratio. OCTA is considered a reliable tool in the detection and quantification of macular ischemia in diabetics.

In this study, the investigators aim to compare the effect of repeated intravitreal injections of ranibizumab and bevacizumab on the perfusion of different capillary layers in the macula of diabetic patients using OCTA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years old with type 1 or 2 diabetes mellitus with decreased BCVA due to center involving diabetic macular edema on spectral-domain optical coherence tomography.
2. Patients with central macular thickness "CMT" of ≥ 300 micrometers

Exclusion Criteria:

1. Ocular conditions that may affect macular perfusion (e.g. retinal vascular diseases, uveitis, vasculitis etc.)
2. History of vitreo-retinal surgeries.
3. Previous macular laser treatment
4. Presence of epi-retinal membrane involving the macula or vitreo-macular traction.
5. Media opacity preventing good image quality.
6. Uncontrolled glaucoma.
7. Thrombo-embolic events within 6 months
8. Previous intravitreal injections of anti-VEGF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in foveal avascular zone area | 0 and 3 months.
  The change in the foveal avascular zone area will be compared between the two treatment arms as a measure of macular perfusion change.
Change in vascular density of the superficial retinal capillary plexus | 0 and 3 months.
  The change in the superficial retinal capillary plexus vascular density will be compared between the two treatment arms as a measure of macular perfusion change.
Change in vascular density of the deep retinal capillary plexus | 0 and 3 months.
  The change in the deep retinal capillary plexus vascular density will be compared between the two treatment arms as a measure of macular perfusion change.

SECONDARY OUTCOMES:
Change in best corrected visual acuity | 0 and 3 months
  The change in best corrected visual acuity will be assessed following treatment with both drugs using standard Snellen charts.
Change in central macular thickness | 0 and 3 months
  The change in central macular thickness will be assessed following treatment with both drugs using optical coherence tomography.
Change in intraocular pressure | 0 and 3 months
  he change in intraocular pressure will be assessed following treatment with both drugs using Goldman applanation tonometry.
Change of severity of diabetic retinopathy | 0 and 3 months
  The change in the severity of diabetic retinopathy will be assessed following treatment with both drugs using color fundus photographs and clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman G Elnahry, MD, PhD, Principal Investigator — Cairo University; Karim M Abdelaty, MBBCH, Study Director — National Eye Center; Ahmed A Abdel-Kader, MD, PhD, Study Chair — Cairo University; Ahmed A Mohalhal, MD, PhD, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michaelides M, Kaines A, Hamilton RD, Fraser-Bell S, Rajendram R, Quhill F, Boos CJ, Xing W, Egan C, Peto T, Bunce C, Leslie RD, Hykin PG. A prospective randomized trial of intravitreal bevacizumab or laser therapy in the management of diabetic macular edema (BOLT study) 12-month data: report 2. Ophthalmology. 2010 Jun;117(6):1078-1086.e2. doi: 10.1016/j.ophtha.2010.03.045. Epub 2010 Apr 22. PMID 20416952
- [Background] Manousaridis K, Talks J. Macular ischaemia: a contraindication for anti-VEGF treatment in retinal vascular disease? Br J Ophthalmol. 2012 Feb;96(2):179-84. doi: 10.1136/bjophthalmol-2011-301087. PMID 22250209
- [Result] Elnahry AG, Abdel-Kader AA, Raafat KA, Elrakhawy K. Evaluation of the Effect of Repeated Intravitreal Bevacizumab Injections on the Macular Microvasculature of a Diabetic Patient Using Optical Coherence Tomography Angiography. Case Rep Ophthalmol Med. 2019 Apr 18;2019:3936168. doi: 10.1155/2019/3936168. eCollection 2019. PMID 31139483
- [Result] Elnahry AG, Abdel-Kader AA, Raafat KA, Elrakhawy K. Evaluation of Changes in Macular Perfusion Detected by Optical Coherence Tomography Angiography following 3 Intravitreal Monthly Bevacizumab Injections for Diabetic Macular Edema in the IMPACT Study. J Ophthalmol. 2020 Apr 27;2020:5814165. doi: 10.1155/2020/5814165. eCollection 2020. PMID 32411431
- [Result] Elnahry AG, Abdel-Kader AA, Habib AE, Elnahry GA, Raafat KA, Elrakhawy K. Review on Recent Trials Evaluating the Effect of Intravitreal Injections of Anti-VEGF Agents on the Macular Perfusion of Diabetic Patients with Diabetic Macular Edema. Rev Recent Clin Trials. 2020;15(3):188-198. doi: 10.2174/1574887115666200519073704. PMID 32427087
- [Result] Elnahry AG, Elnahry GA. Optical Coherence Tomography Angiography of Macular Perfusion Changes after Anti-VEGF Therapy for Diabetic Macular Edema: A Systematic Review. J Diabetes Res. 2021 May 22;2021:6634637. doi: 10.1155/2021/6634637. eCollection 2021. PMID 34124270
- [Result] Elnahry AG, Ramsey DJ. Automated Image Alignment for Comparing Microvascular Changes Detected by Fluorescein Angiography and Optical Coherence Tomography Angiography in Diabetic Retinopathy. Semin Ophthalmol. 2021 Nov 17;36(8):757-764. doi: 10.1080/08820538.2021.1901122. Epub 2021 Mar 30. PMID 33784213
- [Result] Sorour OA, Elsheikh M, Chen S, Elnahry AG, Baumal CR, Pramil V, Abdelhalim TI, Nassar E, Moult EM, Witkin AJ, Duker JS, Waheed NK. Mean macular intercapillary area in eyes with diabetic macular oedema after anti-vascular endothelial growth factor therapy and its association with treatment response. Clin Exp Ophthalmol. 2021 Sep;49(7):714-723. doi: 10.1111/ceo.13966. Epub 2021 Aug 1. PMID 34189816